CLINICAL TRIAL: NCT02456077
Title: Strengthening Physician Communication About HPV Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-2785
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: HPV Immunization Status
Keywords: MCV4: Meningococcal Conjugate Vaccine; HPV: Human Papillomavirus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Practices (Experimental): Intervention offices will adopt a multi-modal vaccine program to increase their patients' vaccine rates.
  Interventions: Behavioral: Multimodal Vaccine Program
- Control Practices (No Intervention): Control offices will offer usual health care related to immunizations throughout the duration of the study.

INTERVENTIONS:
Behavioral: Multimodal Vaccine Program — Efforts will be made to collaborate with pediatric and family medicine offices to utilize a multimodal intervention to improve adolescents' HPV immunization rates. As part of the overall intervention, four intervention strategies will be used: 1) a tailored website, iVac -HPV , 2) Motivational Interview Training for providers, 3) HPV Fact Sheets and 4) The Decision Aid for HPV Vaccines
  Arms: Intervention Practices

SUMMARY:
The purpose of this study is to determine if a multimodal Human Papillomavirus (HPV) immunization program carried out in pediatric and family medicine practices would be more effective in improving adolescent patients' HPV immunization rates than the usual care provided to adolescents in pediatric and family medicine practices.

ELIGIBILITY:
Inclusion Criteria for immunization rate assessment:

1. 9 years of age or older when presenting for care
2. Patients who present for care one year prior to the start of the intervention and up to two years after the start of the intervention

Exclusion Criteria:

1. Less than 9 years of age when presenting for care
2. Patient is not eligible for HPV immunization

Provider survey:

Providers who are working at participating practices during the two times a cross-sectional survey is administered.

Parent survey:

Parents of adolescents who presented for care within one 1 year prior to the two times a cross-sectional survey is administration.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93582 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
The percentage of adolescents who initiate the HPV vaccine series | 1 year
  The percent of eligible patients presenting for care at intervention offices who receive one or more HPV vaccines (using administrative, Electronic Medical Records (EMR), and Colorado Immunization Information System (CIIS) immunization data), during the intervention year, compared to the percent in control offices.

SECONDARY OUTCOMES:
The percentage of adolescents who receive MCV4 vaccine | 1 year
  The percent of eligible patients presenting for care at intervention offices who receive MCV4 vaccine (using administrative, EMR and CIIS immunization data) compared to the percent in control offices.
The percentage of adolescents who receive Tdap vaccine | 1 year
  The percentage of eligible patients presenting for care at intervention offices who receive Tetanus, Diphtheria, Pertussis (Tdap) vaccine (using administrative, EMR and CIIS immunization data) during the intervention year compared to the percent in control offices.
Provider HPV vaccine recommendations | 1 year
  The change in intervention providers' HPV vaccine communication practices compared to control providers' as measured by self-report prior to the intervention and after the intervention.
Parents' experiences and preferences regarding provider communication about HPV vaccines | 1 year
  The change in intervention parents' experiences and preferences regarding provider HPV vaccine communication compared to parents of adolescents attending control practices as measured by self report prior to the intervention and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Dempsey, MD, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Dempsey AF, Pyrznawoski J, Lockhart S, Barnard J, Campagna EJ, Garrett K, Fisher A, Dickinson LM, O'Leary ST. Effect of a Health Care Professional Communication Training Intervention on Adolescent Human Papillomavirus Vaccination: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2018 May 7;172(5):e180016. doi: 10.1001/jamapediatrics.2018.0016. Epub 2018 May 7. PMID 29507952